CLINICAL TRIAL: NCT01872754
Title: Randomized and Single Blind Study Comparing Remifentanil Sedation Versus Propofol for Performing Bronchial Fibroscopies Under Intravenous Anesthesia
Brief Title: Study Comparing the Use of Remifentanil Versus Propofol for Performing Bronchial Fibroscopy
Acronym: REVPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P090803; 2011-005175-17 (Other: IDRCB)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Realisation of Bronchial Fibroscopy
Keywords: Bronchial fibroscopy; Remifentanil; Propofol; Sedation; Target Controlled Infusion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2: Propofol (Active Comparator): Control arm: the use of TCI of hypnotic (Propofol) during realization bronchial fibroscopy.
  Interventions: Drug: 2: Propofol
- 1: Remifentanil (Experimental): Interventional arm: the use of TCI of morphinomimetic (Remifentanil) during realization bronchial fibroscopy.
  Interventions: Drug: 1: Remifentanil

INTERVENTIONS:
Drug: 1: Remifentanil — 1: Remifentanil group The infusion of Remifentanil by TCI begins at distance from the introduction of fiberoptic. The effect site target is 4 ng / ml.- A titration in increments or decrements (respectively increase or decrease of 1 ng / ml effect site concentration) separated by 1 minute intervals until an OAAS score of 4 and respiratory frequency range between 10 and 20 cycles per minute.
  Arms: 1: Remifentanil
Drug: 2: Propofol — 2: Propofol group- The infusion of Propofol by TCI begins at distance from the introduction of fiberoptic. The effect site target is 2,5 ng / ml.- A titration in increments or decrements (respectively increase or decrease of 0.5 mg / ml concentration effect site) separated by 1 minute intervals until an OAAS score of 4 and included respiratory rate between 10 and 20 cycles per minute.
  Arms: 2: Propofol

SUMMARY:
The purpose of this study is to determine whether the use of Target-Controlled Infusion (TCI) of Remifentanil can deliver better conditions for performing bronchial fibroscopy with spontaneous ventilation (decrease the duration of cough) compared to the use of TCI of Propofol.

DETAILED DESCRIPTION:
Patients with an indication of bronchoscopy under sedation with spontaneous ventilation will be prospectively included in the study.

The proposal for inclusion is presented by the anesthetist performing the anesthetic consultation. Consent form and explanatory notes are given to the patient. The patient has a period of reflection of at least 48 hours in the case of a scheduled endoscopy for signing the consent. For urgent cases a period of 24 hours will be accepted. The patient is informed that the proceedings will be recorded to allow the calculation of the total number of coughing episodes and their duration.

* V-1: Inclusion visit in post-interventional care unit.

  * Check the indication of endoscopy and sedation.
  * Verification of inclusion and non-inclusion criteria.
  * Obtention of signed consent from the patient and inclusion in the study.
  * Randomization : The degree of patient anxiety using a visual analogue scale (VAS) and the operator's experience (the number of years of practice) are required for stratification.
  * Collection of epidemiological data
* V0: Bronchial Fibroscopy.

  * Installation of the patient
  * To ensure operator blindness with respect to the type of drug used (remifentanil versus propofol) for the sedation, the tubing and syringe are hidden by a operative drape. The person collecting the data will also blind to the drug used.
  * Oxygen (6l / min) is administred to the patient using a high concentration oxygen mask with an End-tidal CO2.
  * Collection of basic constants (SBP and DBP, HR, RR, SpO2, EtCO2, OAAS score) prior to anesthesia.
  * 5 sprays of lidocaine 50 mg / ml are administred in each nostril.
  * Collection of constants during endoscopy under anesthesia (SBP and DBP, HR, RR, SpO2, EtCO2, OAAS score every minute for the total duration of endoscopy) and the occurrence of cough by sound digital recording. The duration and number of episodes of coughing will be timed retrospectively from the sound recording.
  * Concentration at target effect site is recorded every minute
  * The total dose of lidocaine 10 mg / ml instilled by the operator is recorded. The total dose does not exceed 200 mg.
  * Vital signs (SBP and DBP, HR, RR, SpO2, EtCO2), the total duration of the endoscopy and the number of episodes of coughing by sound recording, OAAS score, the target concentrations at effect site, the type of procedure performed (LBA, biopsies...) and adverse events are collected.
* V1: Visit of end of endoscopy. Satisfaction of the fibroscopist is collected by questionnaire in two areas: the quality of endoscopy in three items (quality of visualization of the tracheobronchial tree, review performance, and ease of progression), and the quality of sedation in three items (interference due to patient movement, coughing related incidents and those linked to the actions of the anesthetist). Each item is measured using a Likert scale of 5 points.
* V2 : Visit of end of study. Patient satisfaction is collected in 3 areas: collecting the degree of inconvenience in three items (pain, memory and cough), the degree of discomfort three items (during local anesthesia, during insertion of the endoscope, and during the exploration of the tracheobronchial tree), and the degree of acceptance to repeat the examination in the future. Each item is measured using a Likert scale of 5 points.
* V3 : patient status. Day 7, patient satisfaction is collected by phone contact or directly if the patient is still in hospital.Patient satisfaction is collected in 3 areas: collecting the degree of inconvenience in three items (pain, memory and cough), the degree of discomfort three items (during insertion of the endoscope, during the exploration of the tracheobronchial tree), and the degree of acceptance to repeat the examination in the future. Each item is measured using a Likert scale of 5 points.
* Effective calculation. We evaluated two strategies for sedation during a preliminary study of 45 patients (Gaillard, SRLF 2010 summary 003940). Cough of more than 10 seconds occurred in 76% of patients sedated with propofol and 32% of patients sedated with Remifentanil. From these data, A number of N = 71 patients will have a power of 80% to demonstrate a difference by Fisher exact probability test between two groups of 35% of percentage of cough of more than 10 secondes.
* Statistical analysis. The primary endpoint and secondary endpoints will be analyzed by qualitative test of Mantel-Haentzel. The homogeneity of odds ratios (existence of a significant level of anxiety) will be tested by the Breslow-Day.Comparing the duration of each examination, the dose of lidocaine instilled, satisfaction scores and the number of increments and decrements in both groups will be made by Mann-Whitney test. For these variables, the possible interactions between the type of action and treatment are analyzed in a ANOVA model.

The duration of recruitment is 45 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient major with consent
* Patient with an indication of bronchoscopy under intravenous sedation:

  * Cough making endoscopy impossible despite local anesthesia
  * Refusal of the patient to undergo the action without sedation
  * There is no limitation related to the type of pathology: it is patient "all comers"

Exclusion Criteria:

* Patients with a known allergy to Remifentanil
* Patients with a known allergy to Propofol, soy, peanuts
* Pregnant women or nursing
* Neurological pathology causing intracranial hypertension
* Patients with a Body Mass Index greater than 30
* Indications of orotracheal intubation :

  * Protection of the upper airways: patient considered "full stomach": Diabetes with autonomic dysfunction, severe gastroesophageal reflux, severe obesity and morbid hiatal hernia and any other situation governed by the anesthesiologist as a situation of full stomach
  * The need for mechanical ventilation severe hypoxemia
* Cirrhosis child B and C
* Intermittent or severe uncontrolled asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Duration of patient's caught | at day0
  Comparison of the duration of patient's caught during realisation of bronchial fibroscopy according to type of performed sedation (remifentanil versus propofol

SECONDARY OUTCOMES:
Respiratory frequence and Gaz volume | Day0
  Compare treatment modalities in terms of side effects (remifentanil versus propofol): initial values, maximum and minimum EtCO2 score, the occurrence of desaturation of more than 3 points compared to baseline in 6 l / min oxygen mask, the occurrence of bradypnea with respiratory rate less than 8 / minute, the occurrence of upper airway obstruction and a inhalation salivary.
Fibroscopist's satisfaction | Day0
  Compare treatment modalities in terms of satisfaction for fibroscopist in 2 areas: the quality of fibroscopy and quality of sedation.
Patient's satisfaction | Day0
  Compare treatment modalities in terms of satisfaction to the patient in 3 areas: collecting the degree of inconvenience, the degree of discomfort and the degree of acceptance to repeat the examination in the future.
Pharmacodynamics | Day0
  Compare treatment modalities in terms pharmacodynamics: target concentrations were collected on initial site effect, maximum and average, as well as the rate received per minute and the total dose.
Number of episodes of cough | Day0
  Compare the number of episodes of cough according to the type of sedation used

CONTACTS AND LOCATIONS:
Overall Officials: Véronique J MAUREL, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint-Louis - Anesthésie Réanimation, Paris, France